CLINICAL TRIAL: NCT04940039
Title: Clinical Study to Assess the Treatment of Schizophrenia With Paliperidone Palmitate in Rwandan Healthcare Settings
Brief Title: A Study to Assess the Treatment of Schizophrenia With Paliperidone Palmitate in Rwandan Healthcare Settings
Acronym: CASPAR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen-Cilag International NV (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR108924; R092670PSY4002 (Other: Janssen-Cilag International NV)
Record Dates: First submitted 2021-06-22; First posted 2021-06-25 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Schizophrenia
Keywords: Long-acting injectable antipsychotics; Low income countries; schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Risperidone; Paliperidone Palmitate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Paliperidone Palmitate (Experimental): Participants in Observation Phase will receive their treatment prescribed by treating physicians as part of their routine clinical practice and the standard of care (SoC) treatment for Rwanda mental healthcare settings. Participants who have not received risperidone or paliperidone or paliperidone palmitate earlier in Observation Phase will receive oral risperidone 3 milligram (mg) tablets once daily for 3 days in Run-in Phase to determine tolerability. Participants will receive flexible dose range from 50 to 150 mg equivalent (eq.) long acting formulation of paliperidone palmitate once monthly (PP1M) as an intramuscular (IM) injection in Lead-in Treatment Phase for at least 17 weeks (maximum 25 weeks) and if stable dose is achieved for PP1M, participants will enter Maintenance Treatment Phase and continue to receive flexible dose range from 175 to 525 mg eq. long acting formulation of paliperidone palmitate every 3 months (PP3M) as an IM injection for up to 24 weeks.
  Interventions: Drug: Risperidone 3 mg; Drug: Paliperidone Palmitate 50 mg eq.; Drug: Paliperidone Palmitate 75 mg eq.; Drug: Paliperidone Palmitate 100 mg eq.; Drug: Paliperidone Palmitate 150 mg eq.; Drug: Paliperidone Palmitate 175 mg eq.; Drug: Paliperidone Palmitate 263 mg eq.; Drug: Paliperidone Palmitate 350 mg eq.; Drug: Paliperidone Palmitate 525 mg eq.

INTERVENTIONS:
Drug: Risperidone 3 mg — Participants will receive 3 mg oral risperidone tablet once daily for 3 days.
Drug: Paliperidone Palmitate 50 mg eq. — Participants will receive 50 mg eq. PP1M IM injection for at least 17 weeks (maximum 25 weeks).
  Other Names: R092670
Drug: Paliperidone Palmitate 75 mg eq. — Participants will receive 75 mg eq. PP1M IM injection for at least 17 weeks.
  Other Names: R092670
Drug: Paliperidone Palmitate 100 mg eq. — Participants will receive 100 mg eq. PP1M IM injection for at least 17 weeks.
  Other Names: R092670
Drug: Paliperidone Palmitate 150 mg eq. — Participants will receive 150 mg eq. PP1M IM injection for at least 17 weeks.
  Other Names: R092670
Drug: Paliperidone Palmitate 175 mg eq. — Participants will receive 175 mg eq. PP3M IM injection up to 24 weeks.
  Other Names: R092670
Drug: Paliperidone Palmitate 263 mg eq. — Participants will receive 263 mg eq. PP3M IM injection up to 24 weeks.
  Other Names: R092670
Drug: Paliperidone Palmitate 350 mg eq. — Participants will receive 350 mg eq. PP3M IM injection up to 24 weeks.
  Other Names: R092670
Drug: Paliperidone Palmitate 525 mg eq. — Participants will receive 525 mg eq. PP3M IM injection up to 24 weeks.
  Other Names: R092670

SUMMARY:
The purpose of this study is to assess the long-term symptomatic response (Visit 2 [Week 1] to Visit 14/Week 66 [End of Study {EOS}]) measured by change in the Clinical Global Impressions -Severity for Schizophrenia (CGI-SS) in participants with schizophrenia who are treated in Rwandan real-world healthcare settings with the antipsychotic regimen that starts with oral anti-psychotic (AP) formulation followed by continued treatment with (paliperidone palmitate 1-month [PP1M] and 3-month [PP3M] formulations).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia by Mini International Neuropsychiatric Interview (MINI)-Screen / MINI (Module K) that requires treatment initiation or a change in treatment to better address safety, efficacy, or adherence limitations of current treatment
* Eligible for treatment in the Rwandan mental healthcare system
* At least moderately ill as measured by the Clinical Global Impression - Severity of Schizophrenia (CGI-SS) scale for schizophrenia (rating of greater than or equal to [>=] 4). This criterion needs to be re-confirmed at Visit 2
* Has a primary caregiver who is willing to participate in this study (caregiver should be knowledgeable about the participant's condition, provide economic/cost of care information, and is expected to be with the participant for greater than [>] 24 hours each week for the duration of the study)
* A woman of childbearing potential must have a negative highly sensitive serum (beta-human chorionic gonadotropin [beta-hCG]) during screening
* Able to give consent to participate in a clinical study that includes treatment with risperidone and long-acting injectable (LAI) formulations of paliperidone palmitate. Participants must be willing to receive injections. The participant and the caregiver must sign their own informed consent form (ICF) indicating that he or she understands the purpose of, and procedures required for, the study and is willing to participate in the study

Exclusion Criteria:

* Has a physical, mental, or legal incapacity that prevents a valid consent or capacity to complete about 12 months of treatment with antipsychotic medication and compliance with this study protocol
* History of organic brain syndromes, comorbid psychiatric and/or physical illnesses, or significant comorbid substance abuse that is likely to interfere with understanding of or compliance with study requirements
* Known allergies, hypersensitivity, or intolerance to risperidone or paliperidone palmitate or its excipients
* Received an investigational intervention including investigational vaccines or used an invasive investigational medical device within 30 days before the planned first dose of study intervention, or is currently enrolled in an investigational study
* Pregnant, or breast-feeding, or planning to become pregnant while enrolled in this study or within 6 months after the last dose of study intervention
* Poor prior response to risperidone or paliperidone

Ages: 19 Years to 34 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 93 (Actual)
Dates: Start 2021-07-22 (Actual); Primary Completion 2024-04-16 (Actual); Study Completion 2024-04-16 (Actual)

PRIMARY OUTCOMES:
Mean Change in Clinical Global Impression Severity of Schizophrenia (CGI-SS) Score from Visit 2 (Week 1) to Visit 14 (Week 66 [End of Study {EOS}]) | Visit 2 (Week 1) to Visit 14 (Week 66 [EOS])
  The CGI-SS will be used to provide a clinical measure of the severity of schizophrenia. It is a single-item Likert scale with a 7-point range (1 indicates none to 7 indicates extreme symptoms).

SECONDARY OUTCOMES:
Mean Change in CGI-SS Score from Visit 6 (Week 25) to Visit 14 (Week 66 [EOS]) | Visit 6 (Week 25) to Visit 14 (Week 66 [EOS])
  The CGI-SS will be used to provide a clinical measure of the severity of schizophrenia. It is a single-item Likert scale with a 7-point range (1 indicates none to 7 indicates extreme symptoms).
Mean Change in CGI-SS Score from Visit 2 (Week 1) to Visit 6 (Week 25) | Visit 2 (Week 1) to Visit 6 (Week 25)
  The CGI-SS will be used to provide a clinical measure of the severity of schizophrenia. It is a single-item Likert scale with a 7-point range (1 indicates none to 7 indicates extreme symptoms).
Change in Personal and Social Performance (PSP) Scale Score from Visit 2 (Week 1) to Visit 14 (Week 66 [EOS]) | Visit 2 (Week 1) to Visit 14 (Week 66 [EOS])
  The PSP scale assesses the degree of difficulty a participant exhibits over a 7-day period within 4 domains of behavior: a) socially useful activities, b) personal and social relationships, c) self-care, and d) disturbing and aggressive behavior. The impairment of each domain is rated on a 6-point basis, including absent (0), mild (1), moderate (2), marked (3), severe (4), and very severe (5). The higher domain score, therefore, indicates, worse functioning in that area.
Change in PSP Scale Scores from Visit 6 (Week 25) to Visit 14 (Week 66 [EOS]) | Visit 6 (Week 25) to Visit 14 (Week 66 [EOS])
  The PSP scale assesses the degree of difficulty a participant exhibits over a 7-day period within 4 domains of behavior: a) socially useful activities, b) personal and social relationships, c) self-care, and d) disturbing and aggressive behavior. The impairment of each domain is rated on a 6-point basis, including absent (0), mild (1), moderate (2), marked (3), severe (4), and very severe (5). The higher domain score, therefore, indicates, worse functioning in that area.
Change in PSP Scale Score from Visit 2 (Week 1) to Visit 6 (Week 25) | Visit 2 (Week 1) to Visit 6 (Week 25)
  The PSP scale assesses the degree of difficulty a participant exhibits over a 7-day period within 4 domains of behavior: a) socially useful activities, b) personal and social relationships, c) self-care, and d) disturbing and aggressive behavior. The impairment of each domain is rated on a 6-point basis, including absent (0), mild (1), moderate (2), marked (3), severe (4), and very severe (5). The higher domain score, therefore, indicates, worse functioning in that area.
Change in Patient Satisfaction Rating Scale Score from Visit 2 (Week 1) to Visit 14 (Week 66 [EOS]) | Visit 2 (Week 1) to Visit 14 (Week 66 [EOS])
  The patient satisfaction rating is a 4-item scale. Two items use a Likert scale with a 6-point range (0 [very dissatisfied] to 5 [very satisfied]) and 2 items are multiple-choice (example, "select all that apply"). Higher score indicates greater satisfaction.
Change in Patient Satisfaction Rating Scale Score from Visit 6 (Week 25) to Visit 14 (Week 66 [EOS]) | Visit 6 (Week 25) to Visit 14 (Week 66 [EOS])
  The patient satisfaction rating is a 4-item scale. Two items use a Likert scale with a 6-point range (0 [very dissatisfied] to 5 [very satisfied]) and 2 items are multiple-choice (example, "select all that apply"). Higher score indicates greater satisfaction.
Change in Patient Satisfaction Rating Scale Score from Visit 2 (Week 1) to Visit 6 (Week 25) | Visit 2 (Week 1) to Visit 6 (Week 25)
  The patient satisfaction rating is a 4-item scale. Two items use a Likert scale with a 6-point range (0 [very dissatisfied] to 5 [very satisfied]) and 2 items are multiple-choice (example, "select all that apply"). Higher score indicates greater satisfaction.
Change in Clinician Satisfaction Rating Scale Score from Visit 2 (Week 1) to Visit 14 (Week 66 [EOS]) | Visit 2 (Week 1) to Visit 14 (Week 66 [EOS])
  The clinician satisfaction rating is a 4-item scale. Two items use a Likert scale with a 6-point range (0 [very dissatisfied] to 5 [very satisfied]) and 2 items are multiple-choice (example, "select all that apply"). Higher score indicates greater satisfaction.
Change in Clinician Satisfaction Rating Scale Score from Visit 6 (Week 25) to Visit 14 (Week 66 [EOS]) | Visit 6 (Week 25) to Visit 14 (Week 66 [EOS])
  The clinician satisfaction rating is a 4-item scale. Two items use a Likert scale with a 6-point range (0 [very dissatisfied] to 5 [very satisfied]) and 2 items are multiple-choice (example, "select all that apply"). Higher score indicates greater satisfaction.
Change in Clinician Satisfaction Rating Scale Score from Visit 2 (Week 1) to Visit 6 (Week 25) | Visit 2 (Week 1) to Visit 6 (Week 25)
  The clinician satisfaction rating is a 4-item scale. Two items use a Likert scale with a 6-point range (0 [very dissatisfied] to 5 [very satisfied]) and 2 items are multiple-choice (example, "select all that apply"). Higher score indicates greater satisfaction.
Change in Schizophrenia Quality of Life Scale (SQLS) Score from Visit 2 (Week 1) to Visit 14 (Week 66 [EOS]) | Visit 2 (Week 1) to Visit 14 (Week 66 [EOS])
  The SQLS has 33 items covering topics such as psychosocial feelings and vitality. Response options are never, rarely, sometimes, often, or always. Scoring algorithms yield a 0 to 100 scale, with higher scores indicating lower quality of life.
Change in SQLS Score from Visit 6 (Week 25) to Visit 14 (Week 66 [EOS]) | Visit 6 (Week 25) to Visit 14 (Week 66 [EOS])
  The SQLS has 33 items covering topics such as psychosocial feelings and vitality. Response options are never, rarely, sometimes, often, or always. Scoring algorithms yield a 0 to 100 scale, with higher scores indicating lower quality of life.
Change in SQLS Score from Visit 2 (Week 1) to Visit 6 (Week 25) | Visit 2 (Week 1) to Visit 6 (Week 25)
  The SQLS has 33 items covering topics such as psychosocial feelings and vitality. Response options are never, rarely, sometimes, often, or always. Scoring algorithms yield a 0 to 100 scale, with higher scores indicating lower quality of life.
Number of Participants with Treatment-emergent Adverse Events | Up to Week 66
  An adverse event is any untoward medical occurrence in a clinical study participants administered a medicinal (investigational or non-investigational) product. An adverse event does not necessarily have a causal relationship with the intervention. Treatment-emergent adverse events are adverse events with onset after the initiation of treatment in observation phase and separately for initiation of paliperidone palmitate (PP) in Lead-in phase or that are a consequence of a pre-existing condition that has worsened after each treatment phase starts.
Number of Participants with Abnormalities in Clinical Laboratory Measures | Up to Week 66
  Number of participants with abnormalities in clinical laboratory measures (including serum chemistry, hematology and urinalysis) will be reported.
Number of Participants with Abnormalities in Vital Signs | Up to Week 66
  Number of participants with abnormalities in vital signs (temperature [oral], pulse/heart rate, and blood pressure) will be reported.
Number of Participants with Abnormalities in Electrocardiogram (ECG) | Up to Week 66
  Number of participants with abnormalities in ECG will be reported.
Number of Participants with Abnormalities in Physical Examination | Up to Week 66
  Number of participants with abnormalities in physical examination (including body weight, waist circumference, and height) will be reported.
Number of Participants With Pregnancy Outcome as a Safety Measure | Up to Week 66
  Number of participants with pregnancy outcome will be reported.
Number of Participants With Suicidal Ideation and Behavior as Assessed by Columbia Suicide Severity Rating Scale (C-SSRS) Score | Visit 12 (Week 46) to Visit 14 (Week 66 [EOS])
  C-SSRS is an approved and standardized scale for the assessment of the severity of suicidality, through clinical interview. The maximum score assigned for each participant will be summarized into one of three categories: no suicidal ideation or behavior (0), suicidal ideation (1-5), suicidal behavior (6-10). Total score ranges from 1 to 10. Higher scores indicate greater severity. Number of participants with suicidal ideation and behavior will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag International NV Clinical Trial, Study Director — Janssen-Cilag International NV
Locations (5):
- Rwanda (5):
  - University Teaching Hospital of Butare(CHUB), Butare
  - Kibuye Referral Hospital, Kibuye
  - CARAES Ndera Neuro-Psychiatric Hospital, Kigali
  - University Teaching Hospital of Kigali, Kigali
  - Rwamagana Provincial Hospital, Rwamagana

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency